CLINICAL TRIAL: NCT01879618
Title: A Phase IIIb Open Label Study To Optimize The Single Bolus Dose Of Dalteparin Sodium For The Prevention Of Clotting Within The Extracorporeal System During Hemodialysis Procedures For Subjects With Chronic Renal Insufficiency: The Parrot Study
Brief Title: Use Of Fragmin In Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6301091
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Chronic Renal Failure
Keywords: Fragmin; dalteparin; hemodialysis; anticoagulation; Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fragmin (Experimental): Fragmin given according to the flexible dosing regimen outlined in the protocol
  Interventions: Drug: Fragmin

INTERVENTIONS:
Drug: Fragmin — variable dosing regimen

SUMMARY:
The study will determine if the Fragmin dose can be adjusted to suit the clinical needs of patients during dialysis.

ELIGIBILITY:
Inclusion Criteria:

* chronic renal failure on hemodialysis

Exclusion Criteria:

* significant comorbidities that would prevent a patient from completing the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Canada (18):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Horizon Health Network/Saint John Regional Hospital, Saint John, New Brunswick
  - Eastern Regional Health Authority, Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Eastern Regional Health Authority, St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - Eastern Regional Health Authority, Waterford Hospital, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Center (QEII) - VG Site, Halifax, Nova Scotia
  - William Osler Health System - Bramptom Civic Hospital, Brampton, Ontario
  - London Health Sciences Centre, University Hospital, London, Ontario
  - London Health Sciences Centre, Kidney Care Centre, London, Ontario
  - William Osler Health System, Orangeville, Ontario
  - Centre intégré de santé et de services sociaux de la Montérégie-Centre, Greenfield Park, Quebec
  - Centre externe de néphrologie CISSS de la Montérégie-Centre, Greenfield Park, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM) - Hopital Saint-Luc, Montreal, Quebec
  - CIUSSS du Nord-de-l'Ile-de-Montreal, Montreal, Quebec
  - CHU de Quebec (Pavillon Hotel-Dieu de Quebec), Québec, Quebec
  - Centre externe de néphrologie CISSS de la Montérégie-Centre, Saint-Lambert, Quebec

REFERENCES:
- [Derived] Soroka S, Agharazii M, Donnelly S, Roy L, Muirhead N, Cournoyer S, MacKinnon M, Pannu N, Barrett B, Madore F, Tennankore K, Wilson JA, Hilton F, Sherman N, Wolter K, Orazem J, Feugere G. An Adjustable Dalteparin Sodium Dose Regimen for the Prevention of Clotting in the Extracorporeal Circuit in Hemodialysis: A Clinical Trial of Safety and Efficacy (the PARROT Study). Can J Kidney Health Dis. 2018 Nov 4;5:2054358118809104. doi: 10.1177/2054358118809104. eCollection 2018. PMID 30542622
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301091&StudyName=Use%20Of%20Fragmin%20In%20Hemodialysis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 12 sites in Canada, 10 of which enrolled participants. A total of 152 participants with chronic renal failure, who had at least 30 previous days of hemodialysis (HD) and had received ≤10,000 IU unfractionated heparin or low molectular weight heparin for anticoagulation during the past month were enrolled in the study.
Pre-assignment Details: The Screening Visit was performed within 9 days preceding first HD session where FRAGMIN was administered. The Final Study Visit took place 5 to 15 days after the final study HD session where the participant was treated with Fragmin (# 20 or the last HD session that was completed, if the partcipant prematurely terminated).
Groups:
- FRAGMIN: Participants were initially administered standard FRAGMIN dose of 5000 IU into the arterial side of the dialyzer and were permitted dose adjustments by increments/decrements of 500 or 1000 IU, for subsequent HD sessions depending upon the outcome of previous HD session and any intervening clinical events since previous HD session.
Period: Overall Study
Arm/Group | FRAGMIN
Started | 152
Completed | 131
Not Completed | 21
Not completed — Does not meet entrance criteria | 1
Not completed — Withdrawal by Subject | 1
Not completed — Surgery;changed schedule; not available | 8
Not completed — Protocol Violation | 6
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set consisted of all participants who received at least one dose of study medication.
Arm/Group | FRAGMIN
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.1 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent of Successful HD Sessions
Description: A successful HD session is defined in terms of efficacy of the drug where the HD session had completed as planned: there was no premature termination due to Grade 3 or 4 clotting or saline flush to prevent the loss of the extracorporeal circuit due to clotting; it was not possible to return the participant's blood or assess the exact extent of clotting. HD sessions which terminated prematurely due to Grade 1 or 2 clotting, safety event, machine failure, or access site displacement were excluded from the analysis. The point estimate and 95% CI were computed based on generalized estimating equation (GEE) model for clustered binomial data.
Time Frame: 20 HD sessions (up to 4 hours)
Population: The Full Analysis Set (FAS) was used for all efficacy analyses which included all participants who received at least one dose of study medication. There were 2776 HD sessions from 151 participants included in the primary analysis.
Measure: Mean (95% Confidence Interval); unit: Percentage of HD Sessions
Arm/Group | FRAGMIN
Number analyzed (Participants) | 151
Percentage of HD Sessions | 99.9 [99.7 to 100]

2. Secondary Outcome: Mean Percent of HD Sessions With an Acceptable Dose
Description: A HD session with an acceptable dose is defined in terms of efficacy of the drug: an HD session for which the dose at the next HD session did not need to be changed due to Grade 3 or 4 clotting, bleeding, access compression time > 10 minutes, or other clinical event. The point estimate and 95% CI were computed based on GEE model for clustered binomial.
Time Frame: 20 HD sessions (up to 4 hours)
Population: FAS was used for all efficacy analyses which included all participants who received at least one dose of study medication. For this endpoint, there were 2630 evaluable HD sessions from 148 participants.
Measure: Mean (95% Confidence Interval); unit: Percentage of HD sessions
Arm/Group | FRAGMIN
Number analyzed (Participants) | 148
Percentage of HD sessions | 89.8 [87.4 to 91.9]

ADVERSE EVENTS:
Time Frame: From screening (-9 days) up to 30 days after last dose of study drug.
Arm/Group | FRAGMIN
Serious Adverse Events (participants affected / at risk) | 3/152
Other Adverse Events (participants affected / at risk) | 27/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FRAGMIN (N=152)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FRAGMIN (N=152)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 19 (19)
Hypotension (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.